CLINICAL TRIAL: NCT01918566
Title: The Role of Endogenous GLP-1 in Regulating Glucose Stimulated Brain Activity
Brief Title: The Role of Endogenous GLP-1 (Glycolipoprotein) in Regulating Glucose Stimulated Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKBB 298/12
Record Dates: First submitted 2013-05-08; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Exploratory Behavior
MeSH Terms: conditions — Exploratory Behavior | interventions — Glucose; Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 300ml tap water (Placebo Comparator): Single intragastric instillation of 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: tap water
- Glucose (Active Comparator): Single intragastric instillation of 75g Glucose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 75g Glucose in 300ml tap water via nasogastric tube
- Glucose plus Lactisole (Active Comparator): Single intragastric instillation of 75g Glucose in 300ml tap water with 450ppm lactisole
  Interventions: Dietary Supplement: Single intragastric instillation of 75g Glucose in 300ml tap water with 450ppm lactisole
- Fructose (Active Comparator): Single intragastric instillation of 25g Fructose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: 25g Fructose in 300ml tap water
- Glucose and Exendin (Active Comparator): Single intragastric instillation of 75g glucose in 300ml tap water with 600pmol/kg/min exendin 9-39
  Interventions: Dietary Supplement: 75g glucose in 300ml tap water with 600pmol/kg/min exendin 9-39
- tap water, lactisole (Sham Comparator): Single intragastric instillation of 300ml tap water with 450ppm lactisole
  Interventions: Dietary Supplement: 300ml tap water with 450ppm lactisole

INTERVENTIONS:
Dietary Supplement: tap water
  Arms: 300ml tap water
Dietary Supplement: Single intragastric instillation of 75g Glucose in 300ml tap water via nasogastric tube
  Arms: Glucose
Dietary Supplement: Single intragastric instillation of 75g Glucose in 300ml tap water with 450ppm lactisole
  Arms: Glucose plus Lactisole
Dietary Supplement: 25g Fructose in 300ml tap water
  Arms: Fructose
Dietary Supplement: 75g glucose in 300ml tap water with 600pmol/kg/min exendin 9-39
  Arms: Glucose and Exendin
Dietary Supplement: 300ml tap water with 450ppm lactisole
  Arms: tap water, lactisole

SUMMARY:
Our objective is to investigate neuro-anatomical correlates of the regulation of energy intake by means of functional MRI. Administration of glucose with and without lactisole and exendin as well as fructose is followed by functional brain MRI, and findings are correlated with serum GLP-1 levels as an endogenous satiety signal in humans.

ELIGIBILITY:
Inclusion Criteria:

* right-handed healthy males, no drugs, non-smoking

Exclusion Criteria:

* drug abuse, smoker, left-handed, claustrophobia

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) in healthy volunteers while they performed a working memory task: changes in cerebral blood flow and blood hormones from baseline to treatment | changes from baseline to one hour after treatment
  Whole brain analysis with a cluster-level threshold was followed by an a priori defined region of interest analysis of the dorsolateral prefrontal cortex including a cluster-level threshold and family-wise error adjustment for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland